CLINICAL TRIAL: NCT06767449
Title: Multi-center Cohort Study to Evaluate the Real-world Efficacy and Safety of Zolbetuximab Plus Chemotherapy in Claudin18.2 Positive, HER2 Negative, Advanced Gastric Cancer
Brief Title: Zolbetuximab Claudin18.2 Positive, HER2 Negative, Advanced Gastric Cancer
Acronym: Zolbetuximab
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Sun Young Rha, PI, Yonsei University
Other Study IDs: 4-2024-1274
Record Dates: First submitted 2024-12-24; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Advanced Gastric Cancer
Keywords: Zolbetuximab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — * Treatment effectiveness in the real world (progression-free survival, overall survival, response rate, etc.)
  * Adverse effects will be evaluated according to the NCI CTCAE v5.0
  * Tissue samples collected before treatment, during treatment, and at disease progression will be analyzed using multiplex IHC to assess PD-L1 expression, MMR gene status, and Claudin18.2. Additionally, NGS testing will be conducted to evaluate the correlation with the treatment response to zolbetuximab.
  * Blood samples will be collected before treatment, during treatment, and after treatment completion to analyze ctDNA, scRNAseq, or immune cell profiling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
* Treatment effectiveness in the real world
* Adverse effects
* Tissue samples collected (multiplex IHC to assess PD-L1 expression, MMR gene status, and Claudin18.2)
* Blood samples collected (ctDNA, scRNAseq, or immune cell profiling)

DETAILED DESCRIPTION:
* Treatment effectiveness in the real world (progression-free survival, overall survival, response rate, etc.)
* Adverse effects will be evaluated according to the NCI CTCAE v5.0
* Tissue samples collected before treatment, during treatment, and at disease progression will be analyzed using multiplex IHC to assess PD-L1 expression, MMR gene status, and Claudin18.2. Additionally, NGS testing will be conducted to evaluate the correlation with the treatment response to zolbetuximab.
* Blood samples will be collected before treatment, during treatment, and after treatment completion to analyze ctDNA, scRNAseq, or immune cell profiling.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 19 years of age at the time of consent.
2. The patient must have histologically confirmed locally advanced, unresectable, or metastatic gastric or gastroesophageal junction adenocarcinoma
3. Patient whose tumor expresses CLDN18.2 in ≥ 75% of tumor cells demonstrating moderate to strong membranous CLDN18 staining as determined by local or central IHC testing.
4. The tumor sample must be HER2-negative (IHC 0, 1+, or IHC 2+/ISH-).
5. The patient must have received Zolbetuximab as a first-line treatment.
6. 1 Patient has ECOG performance status 0 or 1.
7. Patient must meet all of the following criteria based on the locally analyzed laboratory tests collected.

   * Hb ≥8 g/dL (For patients who require a transfusion, it is appropriate if Hb ≥9 g/dL after transfusion)
   * ANC ≥1.0 x 10^9/L
   * Platelet ≥75 x 10^9/L
   * Total bilirubin ≤1.5 x ULN without liver metastasis, or <3.0 x ULN if liver metastasis is present
   * AST or ALT ≤2.5 x ULN without liver metastasis, or ≤5 x ULN if liver metastasis is present
   * Estimated creatinine clearance ≥30 mL/min

Exclusion Criteria:

1. Patient has previously received treatment in a clinical trial of zolbetuximab, or a clinical trial that included zolbetuximab as 1 of the treatment options, even if the patient was not given zolbetuximab
2. History of known or suspected hypersensitivity to Zolbetuximab, other monoclonal antibodies, or components of the used formulations.
3. Patient has received prior systemic chemotherapy for locally advanced unresectable or metastatic gastric or GEJ adenocarcinoma. However, patient may have received either neo-adjuvant or adjuvant chemotherapy, immunotherapy or other systemic anticancer therapies as long as it was completed at least 6 months prior to participation.
4. Patients who have received systemic immunosuppressive therapy, including systemic corticosteroids, within 14 days before enrollment. However, patients using physiological replacement doses of hydrocortisone or its equivalent (maximum hydrocortisone 30 mg/day or prednisone 10 mg/day), those who have received a single dose of systemic corticosteroid, or those who have received systemic corticosteroids as premedication for radiologic contrast agents are allowed.
5. Patient has a complete gastric outlet syndrome or a partial gastric outlet syndrome with persistent/recurrent vomiting
6. Per investigator judgment, patient has significant gastric bleeding and/or untreated gastric ulcers that would exclude the patient from participation per investigator Judgment
7. Patient has any other condition, which, in the opinion of the treating physician, makes the patient unsuitable to receive or tolerate zolbetuximab.

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Treatment effectiveness in the real world (progression-free survival, overall survival, response rate, etc.)
  * Adverse effects will be evaluated according to the NCI CTCAE v5.0
  * Tissue samples collected before treatment, during treatment, and at disease progression will be analyzed using multiplex IHC to assess PD-L1 expression, MMR gene status, and Claudin18.2. Additionally, NGS testing will be conducted to evaluate the correlation with the treatment response to zolbetuximab.
  * Blood samples will be collected before treatment, during treatment, and after treatment completion to analyze ctDNA, scRNAseq, or immune cell profiling.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Treatment effectiveness | 2 year
  Progression-free survival, overall survival, response rate
Number of participants with treatment-related adverse events as assessed by CTCAE V5.0 | 2 year
  Adverse effects will be evaluated according to the NCI CTCAE v5.0
molecular marker Analysis | 2 year
  * Tissue samples collected before treatment, during treatment, and at disease progression will be analyzed using multiplex IHC to assess PD-L1 expression, MMR gene status, and Claudin18.2. Additionally, NGS testing will be conducted to evaluate the correlation with the treatment response to zolbetuximab.
  * Blood samples will be collected before treatment, during treatment, and after treatment completion to analyze ctDNA, scRNAseq, or immune cell profiling.

CONTACTS AND LOCATIONS:
Overall Officials: Sun Young Rha, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Result] Niimi T, Nagashima K, Ward JM, Minoo P, Zimonjic DB, Popescu NC, Kimura S. claudin-18, a novel downstream target gene for the T/EBP/NKX2.1 homeodomain transcription factor, encodes lung- and stomach-specific isoforms through alternative splicing. Mol Cell Biol. 2001 Nov;21(21):7380-90. doi: 10.1128/MCB.21.21.7380-7390.2001. PMID 11585919
- [Result] Gunzel D, Yu AS. Claudins and the modulation of tight junction permeability. Physiol Rev. 2013 Apr;93(2):525-69. doi: 10.1152/physrev.00019.2012. PMID 23589827
- [Result] Sahin U, Koslowski M, Dhaene K, Usener D, Brandenburg G, Seitz G, Huber C, Tureci O. Claudin-18 splice variant 2 is a pan-cancer target suitable for therapeutic antibody development. Clin Cancer Res. 2008 Dec 1;14(23):7624-34. doi: 10.1158/1078-0432.CCR-08-1547. PMID 19047087
- [Result] Lee JH, Kim KS, Kim TJ, Hong SP, Song SY, Chung JB, Park SW. Immunohistochemical analysis of claudin expression in pancreatic cystic tumors. Oncol Rep. 2011 Apr;25(4):971-8. doi: 10.3892/or.2011.1132. Epub 2011 Jan 3. PMID 21206985
- [Result] Woll S, Schlitter AM, Dhaene K, Roller M, Esposito I, Sahin U, Tureci O. Claudin 18.2 is a target for IMAB362 antibody in pancreatic neoplasms. Int J Cancer. 2014 Feb 1;134(3):731-9. doi: 10.1002/ijc.28400. Epub 2013 Sep 16. PMID 23900716
- [Result] Sanada Y, Hirose Y, Osada S, Tanaka Y, Takahashi T, Yamaguchi K, Yoshida K. Immunohistochemical study of claudin 18 involvement in intestinal differentiation during the progression of intraductal papillary mucinous neoplasm. Anticancer Res. 2010 Jul;30(7):2995-3003. PMID 20683045
- [Result] Karanjawala ZE, Illei PB, Ashfaq R, Infante JR, Murphy K, Pandey A, Schulick R, Winter J, Sharma R, Maitra A, Goggins M, Hruban RH. New markers of pancreatic cancer identified through differential gene expression analyses: claudin 18 and annexin A8. Am J Surg Pathol. 2008 Feb;32(2):188-96. doi: 10.1097/PAS.0b013e31815701f3. PMID 18223320
- [Result] Shah MA, Shitara K, Ajani JA, Bang YJ, Enzinger P, Ilson D, Lordick F, Van Cutsem E, Gallego Plazas J, Huang J, Shen L, Oh SC, Sunpaweravong P, Soo Hoo HF, Turk HM, Oh M, Park JW, Moran D, Bhattacharya P, Arozullah A, Xu RH. Zolbetuximab plus CAPOX in CLDN18.2-positive gastric or gastroesophageal junction adenocarcinoma: the randomized, phase 3 GLOW trial. Nat Med. 2023 Aug;29(8):2133-2141. doi: 10.1038/s41591-023-02465-7. Epub 2023 Jul 31. PMID 37524953
- [Result] Shitara K, Lordick F, Bang YJ, Enzinger P, Ilson D, Shah MA, Van Cutsem E, Xu RH, Aprile G, Xu J, Chao J, Pazo-Cid R, Kang YK, Yang J, Moran D, Bhattacharya P, Arozullah A, Park JW, Oh M, Ajani JA. Zolbetuximab plus mFOLFOX6 in patients with CLDN18.2-positive, HER2-negative, untreated, locally advanced unresectable or metastatic gastric or gastro-oesophageal junction adenocarcinoma (SPOTLIGHT): a multicentre, randomised, double-blind, phase 3 trial. Lancet. 2023 May 20;401(10389):1655-1668. doi: 10.1016/S0140-6736(23)00620-7. Epub 2023 Apr 15. PMID 37068504